CLINICAL TRIAL: NCT01134250
Title: Phase Ib/II Study of the Tumour-targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Paclitaxel in Patients With Advanced Solid Tumours
Brief Title: Combination Therapy of F16IL2 and Paclitaxel in Solid Tumour Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16IL2TAXO-05/07; 2007-006457-42 (EudraCT Number)
Record Dates: First submitted 2010-05-25; First posted 2010-05-31 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor; Breast Cancer; Metastatic Melanoma; Non-small Cell Lung Cancer (NSCLC)
Keywords: Interleukin, IL2, F16, monoclonal, antibody, cytokine Paclitaxel, breast cancer,solid tumour; metastatic melanoma, non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- F16IL2 in combination with paclitaxel (Experimental)
  Interventions: Drug: F16IL2 in combination with paclitaxel

INTERVENTIONS:
Drug: F16IL2 in combination with paclitaxel — Intravenous (i.v.) infusions of F16IL2 (Dose escalation: from 5 to 35 MioIU, the dose could be further increased until MTD is reached, following a pharmacokinetic-guided design) on days 1, 8, 15, 29, 36 and 43 over 60 minutes via automated device (perfusor), followed by a 1 hour i.v. infusion of paclitaxel (Dose escalation: from 60 up to 90 mg/m2) on days 1, 8, 15, 29, 36 and 43.
  Patients with objective tumor responses or stable disease will receive additional combination therapy for a maximum of 6 months, or until disease progression, unacceptable toxicity or withdrawal of consent.

SUMMARY:
This Phase Ib/II study is an open label, multicenter study.

The study is divided in two parts:

Phase I: an open-label, dose escalation study of F16IL2 in combination with paclitaxel for patients with solid tumours, bladder cancer, breast cancer, metastatic melanoma, mesothelioma, NSCLC, prostate cancer and sarcoma amenable to taxane therapy.

Phase II: a prospective, single-arm, multicentre study of a fixed dose of F16IL2 in combination with paclitaxel, equivalent to stage 1 of the Simon two-stage phase II design, for patients with metastatic melanoma, breast cancer and NSCLC amenable to taxane therapy.

DETAILED DESCRIPTION:
Breast cancer is a major cause of cancer mortality, second only to lung cancer as a cause of cancer death in women. The five-year survival rate for localized breast cancer has increased from 80 percent in the 1950s to 98 percent today. However, the mortality rate in the most advanced forms remains unsatisfactory. Indeed, the extensive use of mammography within screening programs has led to cancers being detected earlier, when early treatments may be more effective. A greater understanding of the molecular biology and genetic expression of breast cancer has therefore led to new pre-surgical and post-surgical treatments, including hormone modulators and monoclonal antibodies. Many of these agents have led to decreased mortality and disease recurrence.

F16 is a human recombinant antibody fragment in the scFv (single chain Fragment variable) format that is directed against tenascin C, an angiogenesis marker common to most solid tumors independent of the tumor type. ScFv(F16) selectively localizes in tumor tissues in animal models as demonstrated both histologically and during mechanistic studies involving mice transfected with orthotopic human tumours.

IL2, the human cytokine interleukin-2, is a potent stimulator of the immune response. It has a central role in the regulation of T cell responses and effects on other immune cells such as natural killer cells, B cells, monocyte/macrophages and neutrophils (Smith, 1988). IL2 can induce tumor regression through its ability to stimulate a potent cell-mediated immune response in vivo (Rosenberg, 2000).

ELIGIBILITY:
Inclusion Criteria:

For Phase I, cohorts 1 to 8, of the study:

* For patient of Phase I cohort 1, i.e. those patients receiving F16IL2 alone, patients must not be amenable to therapy with paclitaxel/taxanes but must be considered by the Principal Investigator to be suitable candidates for F16IL2 therapy alone.
* Histologically or cytologically confirmed solid cancer with/without evidence of locally advanced or metastatic disease.
* For advanced solid cancer patients, patients may have received previous chemotherapy or radiation therapy, but they must be amenable for paclitaxel treatment according to the discretion of the principal investigator.

For Phase I, cohorts 9 onwards:

* Histologically or cytologically confirmed bladder cancer, breast cancer, unresectable metastatic (stage IV) non-uveal melanoma, mesothelioma, NSCLC, prostate cancer or sarcoma.
* Prior therapies for metastatic disease are allowed, but patients must be amenable for paclitaxel treatment according to the discretion of the principal investigator.
* For breast cancer patients only: patients not suitable for trastuzumab therapy (i.e., no evidence of HER2-overexpressing disease, or trastuzumab therapy exhausted in HER2-overexpressing disease).

For Phase II of the study:

* Histologically or cytologically confirmed breast cancer, unresectable metastatic (stage IV) non-uveal melanoma, or NSCLC.
* Prior therapies for metastatic disease are allowed, but patients must be amenable for paclitaxel treatment according to the discretion of the principal investigator.
* For breast cancer patients only: patients not suitable for trastuzumab therapy (i.e., no evidence of HER2-overexpressing disease, or trastuzumab therapy exhausted in HER2-overexpressing disease).

For phase I and II of the study:

* Patients aged ≥ 18 years.
* Prior radiation therapy is allowed, if the irradiated area is not the only source of measurable or assessable disease.
* ECOG performance status ≤ 2
* Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria (see Section APPENDIX A). This lesion must not have been irradiated during previous treatments.
* All acute toxic effects (excluding alopecia) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v3.0) Grade ≤ 1.
* Sufficient hematologic, liver and renal function:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, haemoglobin (Hb) ≥ 9.5 g/dl.
  * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and or aspartate aminotransferase ≤ 3 x upper limit of reference range (ULN), and total bilirubin ≤ 2.0 mg/gL unless liver involvement by the tumor, in which case the transaminase levels could be up to 5 x ULN.
  * Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 50 mL/min.
* Life expectancy of at least 12 weeks.
* Documented negative test for human immunodeficiency virus.
* Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
* If of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
* Evidence of a personally signed and dated Ethics Committee-approved Informed Consent form indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion criteria:

* For metastatic melanoma patients: Primary ocular melanoma
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, or any cancer curatively treated < 2 years prior to study entry, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, TIs & TI).
* Presence of active infections (e.g. requiring antibiotic therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Presence of known brain metastases. If patient is symptomatic, negative CT scan within two months before study beginning is required. However, presence of controlled brain metastases (i.e., evaluated as SD of PR after radiotherapy) is allowed.
* History of chronic hepatitis B or C, or chronic active hepatitis or active autoimmune diseases.
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
* Irreversible cardiac arrhythmias requiring permanent medication.
* LVEF </= 50% and/or abnormalities observed during baseline MUGA, ECHO or ECG investigations.
* Uncontrolled hypertension.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe rheumatoid arthritis.
* Severe diabetic retinopathy.
* History of allograft or stem cell transplantation.
* Major trauma including surgery within 4 weeks of administration of study treatment.
* Known history of allergy to IL-2, taxanes, or other intravenously administered human proteins/peptides/antibodies.
* Pregnancy or breast feeding. Female patient must agree to use effective contraception, or be surgically sterile or postmenopausal. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Chemotherapy (standard or experimental) within 4 weeks of the administration of study treatment .
* Radiation therapy within 6 weeks of the administration of study treatment.
* Treatment with an investigational study drug within six weeks before beginning of treatment with F16-IL2.
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment.
* Neuropathy > Grade 1.
* The chronic administration of low dose corticosteroids is allowed: however the maximum allowed dose per day cannot exceed 5 mg of prednisone (or equivalent) and it is meant to address cancer symptoms (e.g., pain, dyspnoea, lack of appetite). A suspected presence of chronic inflammatory disease has to be considered an exclusion criterion.
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08-06 (Actual); Primary Completion 2014-04-07 (Actual); Study Completion 2014-04-07 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) and the recommended dose (RD) of F16IL2 when administered in combination with paclitaxel (Phase I). | 28 days
  Safety evaluations performed days 1 through 28, including AEs, SAEs and standard laboratory assessments graded according to the NCI-CTCAE, v3, will be used for determination of dose limiting toxicity (DLT).
To investigate the efficacy of F16IL2, in terms of objective response rate in combination with paclitaxel in metastatic melanoma, breast cancer and NSCLC patients amenable to taxane therapy (Phase II) | 8 weeks
  The primary efficacy endpoint is the proportion of patients achieving a Tumour Response at week 8.

SECONDARY OUTCOMES:
To investigate the safety and tolerability of F16IL2 and paclitaxel when given as a combination (Phase I/II). | 8 weeks
  Safety and tolerability will be assessed through physical examinations, vital signs, laboratory tests (including serum chemistries, hematology parameters) and the recording of adverse events. Treatment emergent adverse events will be summarized by NCI-CTCAE, version 3. Laboratory values and change in vital signs will be summarized.
Investigate pharmacokinetics of F16IL2 and paclitaxel when given as a combination. | 2 weeks
  In order to investigate the PK profile of F16IL2 and paclitaxel, blood samples for PK measurements in serum will be collected at defined time points during weeks 1 and 2 (after the first dose of study drug) in order to assess accumulation of F16IL2/paclitaxel. PK samples will be collected from all patients enrolled in the phase I part of the study (from cohort 9 onwards, pharmacokinetics of F16IL2 only will be performed), and from the first 5 patients in each indication enrolled in the phase II part of the study.
Human anti-fusion protein antibodies | 18 months
  Phase I: To investigate the induction of human anti-fusion protein antibodies (HAFA).
Antitumor activity | 12 months
  To investigate the antitumor activity of the combination of F16IL2 and paclitaxel in solid tumour patients, for cohorts 1 to 8, and in bladder cancer, breast cancer, metastatic melanoma, mesothelioma, non-small cell lung cancer (NSCLC), prostate cancer and sarcoma patients, for cohort 9 onward.
Assessment of median progression-free survival and median overall survival. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Matilde Catania, Dr, Principal Investigator — European Institute of Oncology Milan (Italy)
Locations (5):
- Italy (5):
  - A.O. UNIVERSITARIA OSPEDALI RIUNITI - OSPEDALE UMBERTO I DI ANCONA - ANCONA (AN) (Italy), Ancona
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Meldola (Fc), Meldola
  - European Institute of Oncology, Milan
  - A.O. UNIVERSITARIA POLICLINICO DI MODENA (Italy), Modena
  - Azienda Ospedaliera Universitaria Senese, Siena